CLINICAL TRIAL: NCT02645487
Title: A Phase I Dose-Escalation Study of Stereotactic Radiosurgery for Brain Metastasis Without Whole Brain Radiation
Brief Title: Stereotactic Radiosurgery (SRS) Dose-Escalation Study for Brain Metastasis
Acronym: SRS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Robert Timmerman, Professor, University of Texas Southwestern Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STU 022015-106
Record Dates: First submitted 2015-12-30; First posted 2016-01-01 (Estimated); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Brain Neoplasms, Adult, Malignant
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stereotactic Radiosurgery (Experimental): Radiation, Stereotactic Radiosurgery Dose-Escalation
  Interventions: Radiation: Stereotactic Radiosurgery

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery — Radiation, Stereotactic Radiosurgery Size <= 1cm: 24 Gray (Gy); + 3 Gy incremental escalation up to 30 Gy >1-2cm: 21 Gy; + 3 Gy incremental escalation up to 27 Gy >2-3cm: 18 Gy; + 3 Gy incremental escalation up to 24 Gy
  Other Names: SRS

SUMMARY:
SRS dose escalation for brain metastases in radiation-naïve patients will establish true tolerable doses, which may exceed the current standard doses. This may lead to an improvement in local control, patient survival, and/or quality-of life.

DETAILED DESCRIPTION:
Recently, several large randomized studies have shown that in patients with limited brain metastases, whole brain radiation can be safely deferred when treated with SRS and close surveillance. In light of this, most of such patients are now treated with SRS alone without WBRT. However, the SRS doses set by Radiation Therapy Oncology Group (RTOG) 90-05 continue to be applied to patients without previous cranial irradiation.

The potential insufficiency of current SRS dose for long-term tumor control is of pressing concern. The advances chemotherapy has led to an improvement in overall survival in many patients with metastatic cancer, including malignancies often associated with brain metastases, such as lung (40-50%) and breast (15%). As these patients survive longer, more patients may develop brain metastases and the current dose of SRS may not be adequate to control the brain metastases for the duration of their survival. In fact, there is evidence that the control rate declines with time after SRS, and after 3 years, the local control rate may be only about 60%. In the case of brain metastases from relatively radio-resistant melanoma, the reported 12-months local control rates for SRS range from 52% to 75%. More potent SRS doses could lead to improved long-term control of brain metastases.

ELIGIBILITY:
Inclusion Criteria

1. Biopsy-proven non-hematopoietic malignancy, except for small cell lung cancer, germ cell cancer, or unknown primary tumor.
2. Radiographic evidence by MRI (or by CT scan with CT contrast if ineligible or intolerant of MRI) of brain metastasis. (If patient is unable to tolerate MRI contrast, an MRI without contrast is acceptable if lesions are visible)
3. All brain metastases must be outside the brain stem (midbrain, pons and medulla).
4. Patient must have 10 or less brain metastases.
5. The maximum diameter of any lesion must be less than or equal to 3.0 cm.
6. Previous treatment with surgery, radiation, chemotherapy, immunotherapy or any targeted agents are allowed provided that:

   * Radiation was not to the brain.
   * Surgery to the brain was > 7 days prior to SRS and there remains at least one additional brain metastasis that can be targeted with SRS
7. Age ≥ 18 years.
8. ECOG Performance Score of 2 or better/Karnofsky Performance Status score of 50-60 or better.
9. All men, as well as women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.

   A female of child-bearing potential is any woman (regardless of sexual orientation, marital status, having undergone a tubal ligation, or remaining celibate by choice) who meets the following criteria:
   * Has not undergone a hysterectomy or bilateral oophorectomy; or
   * Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria

1. Patients had craniotomy and surgery to the brain within 7 days from the date of SRS.
2. Patients with leptomeningeal metastasis.

   NOTE: For the purposes of exclusion, LMD is a clinical diagnosis, defined as positive CSF cytology and/or equivocal radiologic or clinical evidence of leptomeningeal involvement. Patients with leptomeningeal symptoms in the setting of leptomeningeal enhancement by imaging (MRI) would be considered to have LMD even in the absence of positive CSF cytology, unless a parenchymal lesion can adequately explain the neurologic symptoms and/or signs. In contrast, an asymptomatic or minimally symptomatic patient with mild or nonspecific leptomeningeal enhancement (MRI) would not be considered to have LMD. In that patient, CSF sampling is not required to formally exclude LMD, but can be performed at the investigator's discretion based on level of clinical suspicion.
3. Patients with a contraindication to both MRI (with or without contrast) and CT scan (with contrast)
4. Patients with life expectancy < 3 months.
5. Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements.
6. Subjects must not be pregnant or nursing at the time of SRS treatment due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Estimated)
Dates: Start 2015-12-18 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Maximal tolerated doses | 90 days
  To identify the maximal tolerated doses for single-fraction stereotactic radiosurgery, within 90 days from the date of procedure, in patients with brain metastases who have not undergone prior brain irradiation.

SECONDARY OUTCOMES:
Overall survival | 3 years
  To evaluate the overall survival (OS), which is defined as the time between date of SRS and the date of death due to any cause.
Time to progression | 3 years
  To evaluate time to progression (TTP), which is defined as the time between date of SRS and date of documented progression. Specific TTP will be determined for the target lesion, non-target lesions, and elsewhere in brain.
Local progression rate | 3 years
  To evaluate the local progression rate of the target lesion. Local progression will be defined by MRI (with or without contrast)/CT (with contrast) imaging according to the modified RECIST 1.1 criteria. Suspected radiation necrosis and/or pseudoprogression will be similarly evaluated
Response rate | 3 years
  To evaluate the response rate, consisting of complete response (CR) and partial response according to the modified RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Timmerman, MD, Principal Investigator — UTSW
Locations (1):
- University of Texas Southwestern Medical Center, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No